CLINICAL TRIAL: NCT03638076
Title: Un-randomized, Open, Multiple-Dose Study to Evaluate the Safety, Antiviral Activity, and Pharmacokinetics of Morphothiadine Mesilate Capsules (GLS4) /Ritonavir Tablets(RTV) in Patients With Chronic Hepatitis B
Brief Title: The Safety, Antiviral Activity, and Pharmacokinetics of Morphothiadine Mesilate Capsules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DGLS4-16-001
Record Dates: First submitted 2018-07-25; First posted 2018-08-20 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLS4 120 mg+ RTV 100mg，bid (Experimental): Patients with chronic HBV infection will receive GLS4 120 mg+ Ritonavir Tablet 100 mg twice daily for 48 weeks.
  Interventions: Drug: GLS4; Drug: RTV
- GLS4 120 mg+ RTV 100mg，tid (Experimental): Patients with chronic HBV infection will receive GLS4 120 mg+ Ritonavir Tablet 100 mg three times daily for 48 weeks .
  Interventions: Drug: GLS4; Drug: RTV

INTERVENTIONS:
Drug: GLS4 — Subject in group A will receive Mesilate Capsule 120mg twice daily. Subject in group B will receive Mesilate Capsule 120mg three times daily.
  Other Names: Morphothiadine Mesilate Capsule
Drug: RTV — Subject in group A will receive Ritonavir tablet 100mg twice daily.Subject in group B will receive Ritonavir tablet 100mg three times daily.
  Other Names: Ritonavir tablet

SUMMARY:
The Safety, Antiviral Activity, and pharmacokinetics of Morphothiadine Mesilate Capsules/Ritonavir Tablets in Patients with Chronic Hepatitis B

DETAILED DESCRIPTION:
Un-randomized, open Multiple-Dose Study to Evaluate the Safety, Antiviral Activity, and pharmacokinetics of Morphothiadine Mesilate Capsules/Ritonavir Tablets in Patients with Chronic Hepatitis B

20 subjects with Chronic Hepatitis B will be enrolled. 10 subjects will be assigned to group A and receive Morphothiadine Mesilate Capsule 120mg and Ritonavir Tablet 100mg twice daily for 48 weeks. 10 subjects will be assigned to group B and receive Morphothiadine Mesilate Capsule 120mg and Ritonavir Tablet 100mg three times daily for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed informed consent form.
2. Positive HBsAg, positive or negative HBeAg, negative immunoglobulin M( if immunoglobulin M is positive, subject should have laboratory report showed that subject had HBsAg or HBV DNA positive more than 6 months) ; Positive HBsAg, positive or negative HBeAg, liver biopsy report showed evidence of chronic HBV infection, in the case of liver biopsy results, the liver biopsy results shall prevail.
3. Subjects who have not received any antiviral treatment; or if Subjects received treatment with interferon/Peg-interferon, or anti-HBV nucleoside drugs, the drugs should be discontinued at least 3 months prior to the screening.
4. For the subject HBeAg is positive, HBV DNA≥1.0×105 IU/mL（PCR）;For the subject HBeAg is negative , HBV DNA≥1.0×104 IU/mL（PCR）
5. 1.3×ULN≤serum alanine aminotransferase(ALT) ≤5×ULN；
6. 18~65 years old,

Exclusion Criteria:

1. Investigator assessed subjects have other clinically significant abnormalities (other than HBV), such as uncontrollable heart disease, gastrointestinal, blood, nervous or other medical disorders, which may interfere with treatment, assessment, or compliance with the protocol;
2. Laboratory results do not comply with the acceptance criteria at screening;
3. People with positive urinalysis(Such as opioids, barbiturates, benzodiazepines, tricyclic antidepressants, phencyclidine, except for there is document proof that urinalysis positive result due to subject use short period or long period of prescription drug or over-the-counter(OTC) drug.
4. Pregnant female or breast-feeding woman.
5. The result of Fibroscan test was conducted within 6 months before screening is showed that fibroscan score 17.5, or Liver tissue test which was conducted within 24 months before screening showed cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
The mean value of HBV DNA decreased from baseline | Prior to dosing and 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44 and 48 weeks after dosing and 7 days after drug withdrawal.
  The mean value of HBV DNA (unit IU/ml) at different time points in each group was lowered compared with baseline.
Adverse events | From the baseline to 7 days after drug withdrawal.
  To assess the safety and tolerability after dosing.

SECONDARY OUTCOMES:
The mean value of serum HBsAg decreased from baseline. | Prior to dosing and 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44 and 48 weeks after dosing and 7 days after drug withdrawal.
  The mean value of serum HBsAg at different time points in each group was lowered compared with baseline.
The mean value of serum HBeAg(if any) decreased from baseline. | Prior to dosing and 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44 and 48 weeks after dosing and 7 days after drug withdrawal.
  The mean value of serum HBeAg (if any) at different time points in each group was lowered compared with baseline.
Cmax | Intensive blood collection after each administration at day1, day7 and 12 weeks, and before the first administration at 2, 4, 8, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44 and 48 week.
  Maximum observed plasma concentration of GLS4 and RTV.
AUC | Intensive blood collection after each administration at day1, day7 and 12 weeks, and before the first administration at 2, 4, 8, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44 and 48 week.
  Area under the plasma concentration-time curve (AUC)
Css_min | Intensive blood collection after each administration at day1, day7 and 12 weeks, and before the first administration at 2, 4, 8, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44 and 48 week.
  The Css_min of GLS4 and RTV.

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No